CLINICAL TRIAL: NCT07240181
Title: Optimization of Inflammatory Bowel Disease Treatment Through Understanding of Gut Virome Heterogeneity and the Potential for Bacteriophage-based Therapy
Brief Title: OPTImization of Inflammatory Bowel Disease Treatment Through Understanding of Gut VIRome Heterogeneity
Acronym: OPTIVIR
Status: Not yet recruiting | Type: Observational
Sponsor: Andreas Munk Petersen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Andreas Munk Petersen, Professor, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Other Study IDs: H-25044017
Record Dates: First submitted 2025-11-14; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: IBD (Inflammatory Bowel Disease); Crohns Disease; Colitis Ulcerative
Keywords: Bacteriophages; Gut virome; Bacteriophage therapy; Fecal virome transplantation; Fecal filtrate transplantation; Gut microbiome imbalances
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Ulcerative colitis (UC): * Confirmed diagnosis of UC for at least 6 months
  * Age ≥ 18 years
  * Stable medical treatment for IBD during the past 3 months
  * Stable lifestyle within the past month (including diet, physical activity, and sleep habits)
  * Verbal and written informed consent
- Crohns disease (CD): * Confirmed diagnosis of CD for at least 6 months
  * Age ≥ 18 years
  * Stable medical treatment for IBD during the past 3 months
  * Stable lifestyle within the past month (including diet, physical activity, and sleep habits)
  * Verbal and written informed consent
- Primary Sclerosing Cholangitis and Inflammatory Bowel Disease (PSC-IBD): * Confirmed diagnosis of PSC-IBD for at least 6 months
  * Age ≥ 18 years
  * Stable medical treatment for PSC-IBD during the past 3 months
  * Stable lifestyle within the past month (including diet, physical activity, and sleep habits)
  * Verbal and written informed consent
- Healthy controls (fecal donors): Donors who are already part of the existing donor program at the Department of Infectious Diseases, Hvidovre Hospital, will serve as healthy controls. Verbal and written informed consent

SUMMARY:
Title: The Role of Good Viruses in Inflammatory Bowel Disease

Background An imbalance in the bacteria in the gut - called gut dysbiosis - is linked to chronic bowel diseases such as Crohn's disease and ulcerative colitis (IBD). A special and more severe form of IBD, called primary sclerosing cholangitis-associated IBD (PSC-IBD), affects both the gut and the bile ducts, and in serious cases can lead to liver failure. There is currently no cure for IBD.

Research suggests that microorganisms in the gut, especially bacteria and viruses called bacteriophages, play an important role in how the disease develops. Treatment with stool from healthy donors, known as fecal microbiota transplantation (FMT), has proven effective against certain infections and has shown promising results in IBD. A newer and possibly safer method is fecal virome transplantation (FVT), where only the virus part (the gut virome) of the stool is used.

Bacteriophages can kill harmful bacteria and help restore balance in the gut, but their use is still experimental. Therefore, we aim to develop a new treatment by growing bacteriophages from healthy individuals in the lab and using them to restore a healthy balance of bacteria and viruses in the gut of patients with IBD.

Purpose of the study The long-term goal of the study is to improve treatment for IBD by gaining a better understanding of differences in the gut virome between IBD patients and healthy people. We also want to explore whether "fermented" bacteriophages from donor stool can be developed into a future bacteriophage-based therapy.

This will be studied using experimental lab setups and animal models. The study will include 10 healthy stool donors and 30 IBD patients (10 with ulcerative colitis, 10 with Crohn's disease, and 10 with PSC-IBD). The study does not involve any treatments - only the collection of biological samples and access to information about your health from your medical record.

ELIGIBILITY:
Inclusion criteria for patients:

* Confirmed diagnosis of UC, CD, or PSC-IBD for at least 6 months
* Age ≥ 18 years
* Stable medical treatment for IBD (and PSC-IBD) within the past 3 months
* Stable lifestyle within the past month (including diet, exercise, and sleep habits)
* Verbal and written informed consent

Exclusion criteria for patients:

* Use of antibiotics within the past 3 months
* Pregnancy or breastfeeding
* Substance abuse or excessive alcohol consumption (according to Danish Health Authority guidelines)
* Other known comorbidities that may affect the gut microbiome (e.g., type 1 diabetes, other autoimmune diseases, cancer, severe obesity, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is a non-interventional trial aiming to examine the virome/bacteriophages from stool samples of patients with IBD (UC, CD, and PSC-IBD) and compare these with healthy controls (fecal donors).
  Study participants The study will include 30 patients with IBD: 10 with ulcerative colitis (UC), 10 with Crohn's disease (CD), and 10 with PSC-IBD. In each subgroup, 5 participants with active disease and 5 in remission will be included (active disease is defined as fecal calprotectin > 250). In addition, 10 fecal donors will be included as healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
To characterize gut bacteriophages and bacteria in patients with IBD and in healthy controls (fecal donors), both as before and after fermentation in bioreactors | 3 years
  16S rRNA gene and metagenome sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Sofie I Halkjær, PhD, Principal Investigator — Hvidovre University Hospital; Torben S Rasmussen, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No